CLINICAL TRIAL: NCT01107821
Title: Negative Pressure Wound Therapy With the Engenex™-Pump and Bio-Dome™ Dressing, an Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/597
Record Dates: First submitted 2010-04-08; First posted 2010-04-21 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Wounds
Keywords: Pressure sores grade III and IV; Traumatic wounds with considerable soft tissue loss; Wounds after necrotizing fasciitis; Abdominal wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Engenex™-pump (Experimental): Negative Pressure Wound Therapy with the Engenex™-pump and Bio-Dome™ Dressing
  Interventions: Device: Engenex™ pump and Bio-Dome™ Wound Dressing

INTERVENTIONS:
Device: Engenex™ pump and Bio-Dome™ Wound Dressing — Engenex™ pump and Bio-Dome™ Wound Dressing is used.

SUMMARY:
Negative pressure wound therapy (NPWT) has become a powerful tool in wound bed preparation of complex wounds and is routinely used in various disciplines, including general surgery and plastic surgery.

NPWT involves the creation of a controlled subatmospheric pressure in the wound bed. The vacuum is generated by a pump and is distributed over the wound bed by a dressing (mostly a foam or gauze sponge). The therapy has several positive effects on the wound bed, such as improved local blood circulation, stimulation of granulation tissue formation and controlled evacuation of wound exudates. Standard negative pressure applied mostly varies between -120 mmHg and -130 mmHg.A new way of applying NPWT is the Engenex™ system using the Bio-Dome™ Wound Dressing, a specially engineered structure that forms a defined space above the surface of the wound. This space will maintain its size and integrity in the presence of negative pressure and wound fluids and thus effectively imposes strain on the underlying tissue. The material properties of the dressing permit moist wound healing while encouraging efficient removal of exudates. The contact material will not absorb fluid. It has been clinically shown that the Bio-Dome™ Wound Dressing is effective at growing granular tissue in the base of a wound at a safe low negative pressure of -75 mmHg, possibly reducing dressing ingrowth into the wound bed to a minimum.

Our intention is to evaluate NPWT by means of the Engenex™ pump and Bio- Dome™ Wound Dressing in 15 patients. Patients with large soft tissue defects will be examined by a plastic surgeon and if suitable for NPWT they will be treated with the Engenex™ NPWT system.

Before starting NPWT wounds will be evaluated and measured (length, width, depth, volume) if possible. Digital photos will be made and wound swabs will be taken for microbiological examination.Dressing changes will be performed twice weekly, on Monday and Thursday or on Tuesday and Friday. At each dressing change a wound will be re-evaluated and measured.

Other parameters to be noted will be, amongst others: pain, comfort, ease of use,material used, time needed for dressing change, etc.

The NPWT treatment will be carried on for maximum three weeks. During this period plastic surgeons will evaluate whether the wound is ready for surgical closure or not.

If surgical closure after 3 weeks is not yet an option possibility exists that NPWT will be continued.

Every wound will be followed up until complete wound healing after surgical closure.

All patients data will be recorded, secured, evaluated and analysed for both medical parameters and health economic parameters.

ELIGIBILITY:
Inclusion Criteria:

Wounds will be assessed by plastic surgeons to evaluate the indication for wound bed preparation. If suitable for NPWT, they will be treated with Engenex® NPWT-system.

* Suitable wounds include:

  * Pressure sores grade III and IV
  * Traumatic wounds with considerable soft tissue loss
  * Wounds after necrotizing fasciitis
  * Abdominal wounds

Exclusion Criteria:

* Impossibility to adhere the polyurethane film to healthy surrounding skin
* Malignancy in the wound
* Untreated osteomyelitis
* Non-enteric and unexplored fistula
* Undebrided wounds with necrotic tissue
* Exposed organs and blood vessels (Always protect vessels, organs, and nerves by covering them with natural tissues or several layers of fine-meshed, non-adherent synthetic material that form a complete barrier.)
* Increased risk of bleeding
* Patient has one or more medical condition(s), diabetes, including renal, hepatic, hematologic, neurologic, or immune disease that in the opinion of the investigator would make the patient inappropriate for this trial
* The plastic surgeon decides that NPWT therapy should be stopped for other reasons than failure of the NPWT therapy
* Less than two weeks of NPWT

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and efficacy of NPWT with Engenex® | at least 2 weeks
  Following parameters are assessed:
  * Adverse Events
  * Wound size/volume and clinical aspects (odour, masceration): clinical evaluation, digital photography
  * Degree of pain, measured by a numeric scale and the use of analgesics at each dressing intervention.
  * Control of Bioburden: Rate of critical colonization and/or infection
    •% of patients with clinical infection requiring systemic antimicrobial therapy
  * Monitoring of subject's comfort with the dressing in situ, evaluated by subject.
  * Ease of use and dressing application and dressing removal, evaluated by health care personnel

SECONDARY OUTCOMES:
To provide instructions for optimal use of Engenex® | at least 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stan Monstrey, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be